CLINICAL TRIAL: NCT03139643
Title: Assessment of the Predictors and Moderators of Behavior Change
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3555E
Record Dates: First submitted 2016-07-29; First posted 2017-05-04 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Dissonance (Experimental): After reading the materials about their chosen behavior, participants will be asked write an essay about their behavior of choice (studying/exercising). For this essay they will be asked to imagine that they have reached their ideal level of academic achievement/fitness, describe what this would look and feel like, and reflect on how this would impact how they view themselves, their relationships, and their day to day life.
  Interventions: Other: Cognitive Dissonance
- Action Planning (Experimental): After reading the materials about their chosen behavior, participants will be asked to make a detailed plan for the following two weeks based on the following items taken from a study by Sniehotta and colleagues (2004): 1) when to complete studying/exercise, 2) where to complete studying/exercise, 3) how to complete studying/exercise (e.g., what types of exercise- cardio, class, etc. or what types of studying activities- reading, taking notes, creating outlines, etc.), and 4) how often to complete studying/exercise. Participants will be given a calendar as an aid to planning their behavior.
  Interventions: Other: Action Planning
- Reflection (Control Condition) (Placebo Comparator): After reading the materials about their chosen behavior, participants will be asked to summarize and reflect on what they read.
  Interventions: Other: Reflection (Control Condition)

INTERVENTIONS:
Other: Cognitive Dissonance — After reading the materials about their chosen behavior, participants will be asked write an essay about their behavior of choice (studying/exercising). For this essay they will be asked to imagine that they have reached their ideal level of academic achievement/fitness, describe what this would look and feel like, and reflect on how this would impact how they view themselves, their relationships, and their day to day life.
  Arms: Cognitive Dissonance
Other: Action Planning — After reading the materials about their chosen behavior, participants will be asked to make a detailed plan for the following two weeks based on the following items taken from a study by Sniehotta and colleagues (2004): 1) when to complete studying/exercise, 2) where to complete studying/exercise, 3) how to complete studying/exercise (e.g., what types of exercise- cardio, class, etc. or what types of studying activities- reading, taking notes, creating outlines, etc.), and 4) how often to complete studying/exercise. Participants will be given a calendar as an aid to planning their behavior.
  Arms: Action Planning
Other: Reflection (Control Condition) — After reading the materials about their chosen behavior, participants will be asked to summarize and reflect on what they read.
  Arms: Reflection (Control Condition)

SUMMARY:
The current study aims to investigate two potential interventions (i.e., cognitive dissonance and action planning) for inducing behavior change for behaviors important to college students-studying and exercise. In addition, this study will investigate factors that may impact behavior change, such as psychological and neuropsychological variables, to better understand how to bridge the intention-behavior gap.

ELIGIBILITY:
Inclusion Criteria:

* Boston University Psychology 101 students at least 18 years of age
* Able to provide informed consent for the study
* Sufficient command of the English language
* Have experience using a computer and mouse

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | Change from baseline to 4 weeks
  Participants who choose to change their exercising behavior will be administer only this outcome measure; therefore, all participants only complete 1 primary outcome measure.
Studying Questionnaire | Change from baseline to 4 weeks
  Participants who choose to change their studying behavior will be administered only this outcome measure; therefore, all participants only complete 1 primary outcome measure.

SECONDARY OUTCOMES:
Distress Intolerance Index | Change from baseline to 4 weeks
  Measure of distress intolerance.
UPPS Impulsive Behavior Scale (UPPS) | Change from baseline to 4 weeks
  Self-report measure of impulsivity.
Penn State Worry Questionnaire (PSWQ) | Change from baseline to 4 weeks
  Self-report measure of worry.
Self-Control Scale (SCS) | Change from baseline to 4 weeks
  Perceived self-control measure.
Delay Discounting Questionnaire | Change from baseline to 4 weeks
  Monetary choice task.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to 4 weeks
  Self-report measure of sleep quality for the past month.
Center for Epidemiological Studies Depression Scale (CES-D) | Change from baseline to 4 weeks
  Self-report measure of depressive symptoms.
Beck Anxiety Inventory (BAI) | Change from baseline to 4 weeks
  Self-report measure of anxiety symptoms experienced in past week.
Generalized Self-Efficacy Scale | Change from baseline to 4 weeks
  Self-report measure of perceived self-efficacy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patten EA, Kredlow MA, Szuhany KL, Keshishian AC, Otto MW. Catching As and Zs: poor sleep quality predicts failures to increase studying time. Sleep Health. 2020 Feb;6(1):15-18. doi: 10.1016/j.sleh.2019.09.001. Epub 2019 Oct 31. PMID 31676201